CLINICAL TRIAL: NCT01719237
Title: Double Blinded Randomized Control Trial Comparing the Onset and Duration of Ultrasound Guided Supraclavicular Nerve Blocks Using Ropivacaine Versus Ropivacaine-Chloroprocaine Mixture
Brief Title: Trial Comparing the Onset and Duration of Ultrasound Guided Supraclavicular Nerve Blocks Using Ropivacaine Versus Ropivacaine-Chloroprocaine Mixture
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of New Mexico (Other)
Collaborators: VA Palo Alto Health Care System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ChloroRopiSCB
Record Dates: First submitted 2012-10-29; First posted 2012-11-01 (Estimated); Results first posted 2022-09-14 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2012-10

CONDITIONS: Pain
Keywords: Onset; Duration; Upper Limb Block; Ultrasound guided supraclavicular block; Ropivacaine; Chloroprocaine
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ropivacine and Cholroprocaine mixture (Active Comparator): 20 ml's of 1% ropivacaine + 10 ml's of 3% 2-chloroprocaine + 0.1 ml of 1 mg/ml epinephrine
  Interventions: Drug: Ropivacine and Chloroprocaine mixture
- Ropivacine only (Sham Comparator): 30 ml syringe with either 20 ml's of 1% ropivacaine + 10 ml's of normal saline + 0.1 ml of 1mg/ml epinephrine
  Interventions: Drug: Ropivacaine only

INTERVENTIONS:
Drug: Ropivacine and Chloroprocaine mixture — Chloroprocaine is added to Ropivacaine
  Arms: Ropivacine and Cholroprocaine mixture
Drug: Ropivacaine only — Ropivacaine diluted with normal saline instead of chloroprocaine
  Arms: Ropivacine only

SUMMARY:
A double blinded randomized controlled trial comparing the onset and duration of the Onset and Duration of Ultrasound Guided Supraclavicular Nerve Blocks Using a long acting local anesthestic (Ropivacaine) with a mixture of a long and short acting local anesthestic (Ropivacaine-Chloroprocaine Mixture).

DETAILED DESCRIPTION:
Patients will be met preoperatively in the pre-anesthesia holding area as is typical for most orthopedic procedures. An attending anesthesiologist will evaluate the patient and planned surgical procedure and determine if the best anesthetic plan includes a supraclavicular brachial plexus block and will ensure that the patient provides informed consent for their anesthetic plan. Patients who will be having a supraclavicular brachial plexus block as part of their anesthetic will be approached for possible inclusion in the study.

The patient's surgical site will be verified by standard time out procedure. Standard monitoring will be placed including pulse oximetry, EKG, and non-invasive blood pressure cuff. A nasal canula will be placed to provide oxygen. The patient may be given midazolam IV up to 0.05 mg/kg as needed for anxiolysis. The supraclavicular brachial plexus block will be performed by either the attending anesthesiologist or a resident physician directly supervised by the attending anesthesiologist using ultrasound guidance.

The randomization envelope will be handed to an anesthesiologist not involved in the patient's care who will fill a 30 ml syringe with either 20 ml's of 1% ropivacaine + 10 ml's of normal saline + 0.1 ml of 1mg/ml epinephrine or 20 ml's of 1% ropivacaine + 10 ml's of 3% 2-chloroprocaine + 0.1 ml of 1 mg/ml epinephrine. The patient and the physicians performing the nerve block and the assessment after the block,will be blinded to the type of local anesthetic injected.

The physician performing the block will use standard aseptic technique and local anesthetic infiltration of the skin. Then, using ultrasound guidance and a 22g Touhy needle, a supraclavicular brachial plexus block will be placed using 25 mls of the study drug. The time of beginning of injection will be recorded. Starting at 10 minutes after injection, motor and sensory exam in the distribution of the ulnar, median, radial and musculocutaneous nerves using pinprick every 3 minutes until motor block and sensory block is complete. As has been used in prior studies, motor scores of 0, 1, and 2 will be used for no motor blockade (0), partial motor blockade (1), and complete motor blockade (2). Similarly, sensory scores will reflect no change in pinprick sensitivity (0), diminished pinprick sensitivity (1), and complete loss of sensitivity to pinprick (2). Being ready for surgical anesthesia will be defined as a score of 2 for sensory testing. Any patient not achieving a score of 2 on the sensory scale by 40 minutes will be considered a failed block. These scores will be recorded every 3 minutes until the block achieves scores of 2 and 2 or until the patient goes to the operating room (OR).

Once in the OR, data will be collected on whether or not the patient experienced pain on incision, required supplemental pain medicine or sedation, or if the patient required general anesthesia and the reason for needing general anesthesia (e.g. patient discomfort, surgeon request, etc). Post-operatively, a motor and sensory exam will again be performed on the patients for whom the nerve block did not achieve scores of 2 and 2 prior to undergoing surgery and on the patients who required general anesthesia. The patient will be given a card as a reminder to write down the time when he/she noticed pain at site of the operation for the first time and separately the time when he/she took pain medication for the first time. The night of the surgery the patient will be contacted over the phone by one of the investigators to ask the time of pain onset and pain medication administration. Additional data regarding the patient age, weight, type of surgery, and sex will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients who will be having a supraclavicular brachial plexus block as part of their anesthetic will be approached for possible inclusion in the study

Exclusion Criteria:

* patients who are pregnant,
* have an ASA status of IV or greater,
* neuropathy,
* a cast or other impediment to performing a motor or sensory exam in the arm and hand,
* patients under the age of 18,
* long term opioid therapy (longer than 1 month),
* history of opioid abuse and pseudocholinesterase deficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-08; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of New Mexico, Albuquerque, New Mexico, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Ropivacaine and Cholroprocaine Mixture: 20 ml's of 1% ropivacaine + 10 ml's of 3% 2-chloroprocaine + 0.1 ml of 1 mg/ml epinephrine
  Ropivacine and Chloroprocaine mixture: Chloroprocaine is added to Ropivacaine
- Ropivacaine Only: 30 ml syringe with either 20 ml's of 1% ropivacaine + 10 ml's of normal saline + 0.1 ml of 1mg/ml epinephrine
  Ropivacaine only: Ropivacaine diluted with normal saline instead of chloroprocaine
Period: Overall Study
Arm/Group | Ropivacaine and Cholroprocaine Mixture | Ropivacaine Only
Started | 30 | 30
Completed | 30 | 29
Not Completed | 0 | 1
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ropivacaine and Cholroprocaine Mixture | Ropivacaine Only | Total
Number analyzed (Participants) | 30 | 29 | 59
Age, Continuous [Mean (Full Range); unit: years] | 50 [23 to 79] | 46 [18 to 71] | 48 [18 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 16 | 30
  Male | 16 | 13 | 29
Region of Enrollment [Number; unit: participants]
  United States | 30 | 29 | 59
Weight (Kg) [Mean (Standard Deviation); unit: kilograms] | 86.4 (20.5) | 80.7 (19) | 83.6 (20.0)
BMI (Kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] | 30.2 (8.7) | 28.0 (5.7) | 29.1 (7.5)

OUTCOME MEASURES:

1. Primary Outcome: Onset of Surgical Anesthesia
Description: Onset of surgical anesthesia is defined as the time after injection of local anesthetic to the time where no sensation of pinprick in the ulnar, median, radial and musculocutaneous nerves
Time Frame: 45 minutes
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Ropivacaine and Cholroprocaine Mixture | Ropivacaine Only
Number analyzed (Participants) | 30 | 29
minutes
  Ulnar-Sensory | 16 [10 to 28] | 22 [13 to 34]
  Median-Sensory | 9 [4 to 16] | 16 [10 to 22]
  Radial-Sensory | 6 [4 to 10] | 10 [7 to 13]
  Musculocutaneous-Sensory | 9 [4 to 10] | 10 [7 to 16]

2. Secondary Outcome: Duration of Analgesia
Description: Time interval between the end of local anestehtic injection and the patient's first report of pain in the surgical site after surgery
Time Frame: 72 hours
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Ropivacaine and Cholroprocaine Mixture | Ropivacaine Only
Number analyzed (Participants) | 30 | 29
minutes | 566 [428 to 670] | 718 [597 to 851]

ADVERSE EVENTS:
Arm/Group | Ropivacaine and Cholroprocaine Mixture | Ropivacaine Only
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/29
Other Adverse Events (participants affected / at risk) | 4/30 | 1/29
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ropivacaine and Cholroprocaine Mixture (N=30) | Ropivacaine Only (N=29)
Block Failure (Injury, poisoning and procedural complications) | 4 (4) | 1 (1) — Failure of nerve block procedure to provide complete surgical anesthesia

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes